CLINICAL TRIAL: NCT06026813
Title: Pressure Alternating Shoes (PAS) for Prevention of Diabetic Foot Ulcers
Brief Title: Pressure Alternating Shoes
Acronym: PAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH); The University of Texas at Arlington (Other)
Responsible Party: Principal Investigator, Peter Crisologo, DPM, Professor, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STU-2022-1038; 7R21AG061471-02 (NIH)
Record Dates: First submitted 2023-08-25; First posted 2023-09-07 (Actual); Results first posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Foot Ulcer, Diabetic
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Healthy controls (Experimental): Patients without diabetes who do not have foot wounds or history of amputation
  Interventions: Device: test pressure alternating shoes
- Patients with Diabetic Neuropathy (Experimental): Patients with diagnosed diabetes and neuropathy who do not have foot wounds or history of amputation.
  Interventions: Device: test pressure alternating shoes

INTERVENTIONS:
Device: test pressure alternating shoes — test pressure alternating shoes

SUMMARY:
The project is designed to develop and test Pressure Alternating Shoes (PAS), which will periodically off-load certain regions of the foot in order to prevent foot ulcers. An automated dual layer insole compromised of an active pressurized actuator array in combination with a passive compliant layer on top of each actuator to modulate and distribute the plantar surface pressure as desired will be tested. This device will allow us to simultaneously load and offload select areas of the foot using the active layer by inflating and deflating individual actuators using pressurized air. After offloading, the remaining load will be distributed to other areas with inflated actuators. Automatic modulation will be provided through programmable control hardware which will cyclically relieve mechanical loading based on a prescribed duration and frequency.

DETAILED DESCRIPTION:
The two-tier human subjects study will be conducted to assess the biomechanical characteristics of PAS. In the first tier, we will test PAS in healthy subjects and in the second tier, we will test PAS in Diabetic Neuropathy patients (DN).

Subjects will walk on a treadmill in their usual daily shoes for 5 minutes, then with standard diabetic shoes with the PAS insoles for 5 minutes. Subjects will wear body worn sensors that assess position of the body. Subjects will have the temperature of their feet measured via a special camera after walking. Subjects will rest for 30 minute washout period and have the blood flow in the soles of the feet measured via a special camera. 1 healthy subject will undergo MRI of the foot and ankle.

ELIGIBILITY:
Healthy Controls:

Inclusion Criteria:

* Age 18 or greater
* Ability to wear insoles in shoes provided
* Ability to walk unaided

Exclusion Criteria:

* Diabetic Neuropathy
* Charcot foot
* Knee pain
* Previous amputations
* Inflammatory diseases such as rheumatoid arthritis
* Open wounds, ulcers, sores or blisters on the feet; signs of infection in the feet

Diabetic population:

Inclusion:

* Age 18 or greater
* Ability to wear insoles in shoes provided
* Ability to walk unaided
* Diagnosis of diabetic neuropathy

Excluision:

* Charcot foot
* Knee Pain
* Previous amputations
* Inflammatory diseases such as rheumatoid arthritis
* Open wounds, ulcers, sores or blistesr on the feet; signs of infection in the feet

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2024-03-07 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Crisologo, D.P.M., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to design & device constraints, unable to randomize between left/right foot (PAS device) between subjects & were asked to walk with daily shoes on treadmill-5 mins (Control data). Order of sessions (PAS & Daily footwear) weren't randomized as in crossover study. After testing PAS device, daily footwear use data was collected in healthy subjects (Tier 1). Study procedures (use of PAS and daily footwear) in Tier 2- diabetic neuropathic subjects followed the same sequence as in Tier 1.
Groups:
- Healthy Controls (Tier 1): Patients without diabetes who do not have foot wounds or history of amputation.
  Pressure alternating shoe insoles were placed in both the right and left post-operative shoes. Both insoles were inflated to the same pressure to prevent uneven foot elevation and promote stabilization. However, only the right-side insole was connected to the control box to inflate and offload air cells during the test. Due to design and device constraints, we were unable to randomize between the left or right foot between subjects. Although the protocol mentions diabetic footwear, this is a broad phrase that encompasses post operative shoes as there are many real-world patients who use post operative shoes as their footwear. Subjects were then asked to walk with their daily shoes on the treadmill for 5 minutes (Control data). The order of these sessions / sequence (PAS and Daily footwear) were not randomized as in a cross-over study. After testing PAS device, daily footwear (control data) was collected in health subjects (Tier 1). No amendment to the protocol was made for the change in study flow. This was a minor deviation, and we have completed a deviation form for the same and filed it within the study binder.
- Patients With Diabetic Neuropathy (Tier 2): Patients with diagnosed diabetes and neuropathy with superficial ulcers and/or history of surgery/partial amputation.
  Pressure alternating shoe insoles were placed in both the right and left post-operative shoes. Both insoles were inflated to the same pressure to prevent uneven foot elevation and promote stabilization. However, only the right-side insole was connected to the control box to inflate and offload air cells during the test (5 mins). Due to design and device constraints, we were unable to randomize between the left or right foot between subjects. Subjects were then asked to walk with their daily shoes on the treadmill for 5 minutes (Control data). The order of these sessions / sequence (PAS and Daily footwear) were not randomized as in a cross-over study. After testing PAS device, daily footwear (control data) was collected in diabetic neuropathic subjects (Tier 2). No amendment to the protocol was made for the change in study flow. This was a minor deviation, and we have completed a deviation form for the same and filed it within the study binder.
Period: Session 1- Tier 1 Subjects(5 Mins)
Arm/Group | Healthy Controls (Tier 1) | Patients With Diabetic Neuropathy (Tier 2)
Started | 20 | 0
Completed | 20 | 0
Not Completed | 0 | 0
Period: Session 2-Tier 2 Subjects(5 Mins)
Arm/Group | Healthy Controls (Tier 1) | Patients With Diabetic Neuropathy (Tier 2)
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthy Controls- Tier 1: Pressure alternating shoe insoles were placed in both the right and left post-operative shoes. Both insoles were inflated to the same pressure to prevent uneven foot elevation and promote stabilization. However, only the right-side insole was connected to the control box to inflate and offload air cells during the test. Due to design and device constraints, we were unable to randomize between the left or right foot between subjects. Although the protocol mentions diabetic footwear, this is a broad phrase that encompasses post operative shoes as there are many real-world patients who use post operative shoes as their footwear. Subjects were then asked to walk with their daily shoes on the treadmill for 5 minutes (Control data). The order of these sessions / sequence (PAS and Daily footwear) were not randomized as in a cross-over study. After testing PAS device, daily footwear (control data) was collected in health subjects (Tier 1). No amendment to the protocol was made for the change in study flow. This was a minor deviation, and we have completed a deviation form for the same and filed it within the study binder.
- Patients With Diabetic Neuropathy- Tier 2: Patients with diagnosed diabetes and neuropathy with superficial ulcers and/or history of surgery/partial amputation.
  Pressure alternating shoe insoles were placed in both the right and left post-operative shoes. Both insoles were inflated to the same pressure to prevent uneven foot elevation and promote stabilization. However, only the right-side insole was connected to the control box to inflate and offload air cells during the test (5 mins). Due to design and device constraints, we were unable to randomize between the left or right foot between subjects. Subjects were then asked to walk with their daily shoes on the treadmill for 5 minutes (Control data). The order of these sessions / sequence (PAS and Daily footwear) were not randomized as in a cross-over study. After testing PAS device, daily footwear (control data) was collected in diabetic neuropathic subjects (Tier 2). No amendment to the protocol was made for the change in study flow. This was a minor deviation, and we have completed a deviation form for the same and filed it within the study binder.
- Total: Total of all reporting groups
Arm/Group | Healthy Controls- Tier 1 | Patients With Diabetic Neuropathy- Tier 2 | Total
Number analyzed (Participants) | 20 | 1 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 1 | 21
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 17 | 0 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 0 | 5
  Not Hispanic or Latino | 15 | 1 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4 | 0 | 4
  Caucasian | 15 | 0 | 15
  African-American | 1 | 0 | 1
  Black | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Average Pressure at Baseline With Pressure Alternating Shoes, Right Foot (Before Any Cells Were Offloaded)
Description: Maximum Average pressure values in the plantar regions before offloading during walking. The insole consists of seven air cells that align with specific regions: the big toe (cell 1), the area spanning from the second toe to the fifth toe (cell 2), metatarsal heads (cells 3 and 4), the midfoot (cells 5 and 6), and the heel (cell 7). Measurements were only obtained from the right foot.
Time Frame: Before any cells were offloaded (First 40-seconds of the walk)
Population: Due to technical issues like unexpected stop in the interface pressure data collection during testing and insole control box not functioning properly, resulted in incomplete data collection for 4 healthy subjects and therefore not included in the analysis of this outcome measure. All successfully collected data are reported.
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Healthy Controls | Patients With Diabetic Neuropathy
Number analyzed (Participants) | 16 | 1
kPa
  Cell 1 | 118.5 (26.4) | 113.7
  Cell 3 | 96.6 (30.2) | 54.9
  Cell 4 | 83.8 (20.0) | 72.2
  Cell 7 | 95.2 (19.0) | 92.1

2. Primary Outcome: Maximum Average Pressure at After Offloading - Diabetic Footwear Equipped With PAS Device
Description: Maximum Average pressure values in the plantar regions after offloading cells during walking. The insole consists of seven air cells that align with specific regions: the big toe (cell 1), the area spanning from the second toe to the fifth toe (cell 2), metatarsal heads (cells 3 and 4), the midfoot (cells 5 and 6), and the heel (cell 7). Measurements were only obtained from the right foot. The results reported represent results for footwear with PAS device.
Time Frame: After offloading (approx. 41- 200 seconds walk)
Population: Due to technical issues like unexpected stop in the interface pressure data collection during testing and insole control box not functioning properly, resulted in incomplete data collection for 4 healthy subjects and therefore not included in the analysis of this outcome measure. All successfully collected data are reported. This outcome was only assessed for subjects (in both Tiers) with Diabetic Footwear Equipped With PAS Device.
Measure: Mean (Standard Deviation); unit: kPa
Groups:
- Healthy Controls - Footwear With PAS Device: Patients without diabetes who do not have foot wounds or history of amputation
- Patients With Diabetic Neuropathy - Footwear With PAS Device: Patients with diagnosed diabetes and neuropathy who do not have foot wounds or history of amputation.
Arm/Group | Healthy Controls - Footwear With PAS Device | Patients With Diabetic Neuropathy - Footwear With PAS Device
Number analyzed (Participants) | 16 | 1
kPa
  Cell 1 | 97.6 (25.7) | 94.6
  Cell 3 | 82.5 (26.5) | 48.4
  Cell 4 | 70.2 (18.1) | 56.6
  Cell 7 | 83.2 (17.3) | 78.8

3. Primary Outcome: Peak Interface Pressure at Baseline (Before Offloading) - Diabetic Footwear Equipped With PAS Device
Description: Peak Interface Pressure values in the plantar regions before offloading during walking. The insole consists of seven air cells that align with specific regions: the big toe (cell 1), the area spanning from the second toe to the fifth toe (cell 2), metatarsal heads (cells 3 and 4), the midfoot (cells 5 and 6), and the heel (cell 7). Measurements were only obtained from the right foot. The results reported represent results for footwear with PAS device.
Time Frame: Baseline (First 40-seconds of the walk)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Healthy Controls - Footwear With PAS Device | Patients With Diabetic Neuropathy - Footwear With PAS Device
Number analyzed (Participants) | 16 | 1
kPa
  Cell 1 | 146.6 (28.4) | 101.8
  Cell 3 | 125.1 (37.5) | 51.2
  Cell 4 | 98.78 (17.3) | 64.2
  Cell 7 | 107.6 (20.5) | 78.3

4. Primary Outcome: Peak Interface Pressure at After Offloading - Diabetic Footwear Equipped With PAS Device
Description: Peak Interface Pressure values in the plantar regions after offloading during walking. The insole consists of seven air cells that align with specific regions: the big toe (cell 1), the area spanning from the second toe to the fifth toe (cell 2), metatarsal heads (cells 3 and 4), the midfoot (cells 5 and 6), and the heel (cell 7). Measurements were only obtained from the right foot. The results reported represent results for footwear with PAS device.
Time Frame: After offloading (approx. 41- 200 seconds walk)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Healthy Controls - Footwear With PAS Device | Patients With Diabetic Neuropathy - Footwear With PAS Device
Number analyzed (Participants) | 16 | 1
kPa
  Cell 1 | 119.5 (26.32) | 85.6
  Cell 3 | 105.2 (32.3) | 44.7
  Cell 4 | 84.21 (16.4) | 51.7
  Cell 7 | 94.81 (18.8) | 64.1

5. Primary Outcome: Max Average Pressure Change Among All Participants - Diabetic Footwear Equipped With PAS Device
Description: Percentage change due to offloading for each participant is measured by dividing the pressure difference between the after offloading and before offloading values divided by the before offloading value. Measurements were only obtained from the right foot. The results reported represent results for footwear with PAS device.
Time Frame: Baseline (first 40-second walk), 201 seconds after the intervention ended
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Healthy Controls - Footwear With PAS Device | Patients With Diabetic Neuropathy - Footwear With PAS Device
Number analyzed (Participants) | 16 | 1
percent change
  Cell 1 | 18.1 (10.4) | 16.7
  Cell 3 | 14.4 (6.5) | 11.8
  Cell 4 | 16.4 (6.1) | 21.6
  Cell 7 | 12.8 (3.4) | 14.4

6. Primary Outcome: Peak Pressure Change Among All Participants - Diabetic Footwear Equipped With PAS Device
Description: Peak pressure change due to offloading for each participant is measured by dividing the pressure difference between the peak after offloading and peak before offloading values divided by the peak before offloading value. Measurements were only obtained from the right foot. The results reported represent results for footwear with PAS device.
Time Frame: Baseline (first 40-second walk), 201 seconds after the intervention ended
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Healthy Controls - Footwear With PAS Device | Patients With Diabetic Neuropathy - Footwear With PAS Device
Number analyzed (Participants) | 16 | 1
percent change
  Cell 1 | 18.5 (9.3) | 15.9
  Cell 3 | 15.93 (6.1) | 12.6
  Cell 4 | 14.67 (6.8) | 19.5
  Cell 7 | 11.83 (4.8) | 18.0

7. Secondary Outcome: Plantar Skin Temperature at Baseline, Right Foot
Description: Plantar skin temperature measured by a noncontact thermal imaging camera (*Celcius) before the intervention and without footwear
Time Frame: Baseline before the intervention (30 minutes after start of visit 1)
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Healthy Controls | Patients With Diabetic Neuropathy
Number analyzed (Participants) | 20 | 1
degree Celsius
  Right foot | 29.64 (2.16) | 34.7
  Left foot | 29.73 (2.07) | 35

8. Secondary Outcome: Plantar Skin Temperature Post Intervention, Right Foot
Description: Plantar skin temperature measured by a noncontact thermal imaging camera (*Celcius) post intervention, without footwear
Time Frame: Post intervention (215 seconds)
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Healthy Controls | Patients With Diabetic Neuropathy
Number analyzed (Participants) | 20 | 1
degree Celsius
  Right foot | 28.7 (2.04) | 32.1
  Left foot | 29.35 (1.62) | 32.2

9. Secondary Outcome: Tissue Oxygenation (Oxygen Saturation) - for Plantar Lateral Foot
Description: Plantar foot tissue oxygenation (Oxygen saturation) is measured by noncontact hyperspectral imaging camera (StO2). Only the right foot was analyzed and without footwear.
Time Frame: Baseline (30 minutes after start of visit 1)
Population: We gathered and assessed measurements of the plantar lateral foot at baseline for both healthy and diabetic participants combined that is reported here.
Measure: Median (Inter-Quartile Range); unit: percentage StO2
Groups:
- Overall Subjects in Experimental Group: Patients (healthy+ ones with Diabetic Neuropathy) who underwent intervention (test pressure alternating shoes)
Arm/Group | Overall Subjects in Experimental Group
Number analyzed (Participants) | 21
percentage StO2 | 67.0 [64.0 to 72.3]

10. Secondary Outcome: Tissue Oxygenation (Oxyhemoglobin and Deoxyhemoglobin ) - for Plantar Lateral Foot
Description: Plantar foot tissue oxygenation (Oxyhemoglobin and Deoxyhemoglobin) is measured by noncontact hyperspectral imaging (HSI) camera. Only the right foot was analyzed and without footwear. The accepted measure of oxyhemoglobin and deoxyhemoglobin is arbitrary units (AU). NIR spectrum light passes through skin and is reflected off the blood supplying the tissue. Wavelength dependent light absorption of hemoglobin differs if it is carrying oxygen or not, therefore detecting oxygenated and deoxygenated blood. This was derived from Beer-Lambert Law but would need to be verified by the manufacturer. There is no researcher drawn calculation as the device provides the arbitrary unit based on the reflectance detected back to the imaging device. No reference values or any standardization available but one would infer higher oxyhemoglobin level indicates better oxygenation and thus a higher deoxyhemoglobin would be indicative of poor oxygenation.
Time Frame: Baseline (30 minutes after start of visit 1)
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: Arbitrary Units (AU)
Arm/Group | Overall Subjects in Experimental Group
Number analyzed (Participants) | 21
Arbitrary Units (AU)
  Oxyhemoglobin | 0.50 [0.43 to 0.54]
  Deoxyhemoglobin | 0.24 [0.20 to 0.25]

11. Secondary Outcome: Tissue Oxygenation (Oxygen Saturation) - for Plantar Medial Foot
Description: Plantar Medial foot tissue oxygenation (Oxygen saturation) is measured by noncontact hyperspectral imaging camera (StO2). Only the right foot was analyzed and without footwear.
Time Frame: Baseline (30 minutes after start of visit 1)
Population: We gathered and assessed measurements of the plantar medial foot at baseline for both healthy and diabetic participants combined that is reported here.
Measure: Median (Inter-Quartile Range); unit: percentage StO2
Arm/Group | Overall Subjects in Experimental Group
Number analyzed (Participants) | 21
percentage StO2 | 71.0 [66.8 to 72.5]

12. Secondary Outcome: Tissue Oxygenation (Oxyhemoglobin and Deoxyhemoglobin) - for Plantar Medial Foot
Description: Plantar medial foot tissue oxygenation (Oxyhemoglobin and Deoxyhemoglobin) is measured by noncontact hyperspectral imaging (HSI) camera. Only the right foot was analyzed. Only the right foot was analyzed and without footwear. The accepted measure of oxyhemoglobin and deoxyhemoglobin is arbitrary units (AU). NIR spectrum light passes through skin and is reflected off the blood supplying the tissue. Wavelength dependent light absorption of hemoglobin differs if it is carrying oxygen or not, therefore detecting oxygenated and deoxygenated blood. This was derived from Beer-Lambert Law but would need to be verified by the manufacturer. There is no researcher drawn calculation as the device provides the arbitrary unit based on the reflectance detected back to the imaging device. No reference values or any standardization available but one would infer higher oxyhemoglobin level indicates better oxygenation and thus a higher deoxyhemoglobin would be indicative of poor oxygenation.
Time Frame: Baseline (30 minutes after start of visit 1)
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: Arbitrary Units (AU)
Arm/Group | Overall Subjects in Experimental Group
Number analyzed (Participants) | 21
Arbitrary Units (AU)
  Oxyhemoglobin | 0.46 [0.41 to 0.49]
  Deoxyhemoglobin | 0.19 [0.17 to 0.21]

13. Secondary Outcome: Tissue Oxygenation (Oxygen Saturation) - for Plantar Lateral Foot
Description: as for outcome 9
Time Frame: Post Gait (approx. 2015 seconds post intervention)
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: percentage StO2
Arm/Group | Overall Subjects in Experimental Group
Number analyzed (Participants) | 21
percentage StO2 | 71.0 [65.3 to 73.8]

14. Secondary Outcome: Tissue Oxygenation (Oxyhemoglobin and Deoxyhemoglobin ) - for Plantar Lateral Foot
Description: as for outcome 10
Time Frame: Post Gait (approx. 2015 seconds post intervention)
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: Arbitrary Units (AU)
Arm/Group | Overall Subjects in Experimental Group
Number analyzed (Participants) | 21
Arbitrary Units (AU)
  Oxyhemoglobin | 0.50 [0.42 to 0.59]
  Deoxyhemoglobin | 0.21 [0.18 to 0.24]

15. Secondary Outcome: Tissue Oxygenation (Oxygen Saturation) - for Plantar Medial Foot
Description: as for outcome 11
Time Frame: Post Gait (approx. 2015 seconds post intervention)
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: percentage StO2
Arm/Group | Overall Subjects in Experimental Group
Number analyzed (Participants) | 21
percentage StO2 | 73.5 [67.3 to 76.0]

16. Secondary Outcome: Tissue Oxygenation (Oxyhemoglobin and Deoxyhemoglobin) - for Plantar Medial Foot
Description: Plantar medial foot tissue oxygenation (Oxyhemoglobin and Deoxyhemoglobin) is measured by noncontact hyperspectral imaging (HSI) camera. Only the right foot was analyzed and without footwear. The accepted measure of oxyhemoglobin and deoxyhemoglobin is arbitrary units (AU). NIR spectrum light passes through skin and is reflected off the blood supplying the tissue. Wavelength dependent light absorption of hemoglobin differs if it is carrying oxygen or not, therefore detecting oxygenated and deoxygenated blood. This was derived from Beer-Lambert Law but would need to be verified by the manufacturer. There is no researcher drawn calculation as the device provides the arbitrary unit based on the reflectance detected back to the imaging device. No reference values or any standardization available but one would infer higher oxyhemoglobin level indicates better oxygenation and thus a higher deoxyhemoglobin would be indicative of poor oxygenation.
Time Frame: Post Gait (approx. 2015 seconds post intervention)
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: Arbitrary Units (AU)
Arm/Group | Overall Subjects in Experimental Group
Number analyzed (Participants) | 21
Arbitrary Units (AU)
  Oxyhemoglobin | 0.47 [0.38 to 0.52]
  Deoxyhemoglobin | 0.18 [0.15 to 0.21]

17. Secondary Outcome: Balance
Description: Positional sense measured by body-worn sensors (cm)
Time Frame: Baseline
Population: Data were not able to be collected and were considered invalid due to an equipment malfunction (technical difficulties with the sensors).Therefore, this technical issue prevented an assessment and collection of the data.
Arm/Group | Healthy Controls | Patients With Diabetic Neuropathy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: approximately 2 hours
Description: The arms are represented in this fashion to show there were no adverse events between patients with and without diabetic neuropathy as they both received the intervention.
Arm/Group | Healthy Controls | Patients With Diabetic Neuropathy
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/1
Other Adverse Events (participants affected / at risk) | 0/20 | 0/1

LIMITATIONS AND CAVEATS:
Ex-PI left institution after enrollment completion in study. Data not collected for 'Balance' outcome due to technical issues involving body worn sensor connectivity. For remaining, outcomes due to technical issues like unexpected stop in interface pressure data collection during testing & insole control box not functioning properly, it resulted in inability to collect pressure data for 4 healthy subjects & so not included in analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-11-10): https://cdn.clinicaltrials.gov/large-docs/13/NCT06026813/Prot_SAP_001.pdf
  • Informed Consent Form (2024-06-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT06026813/ICF_000.pdf